CLINICAL TRIAL: NCT00949702
Title: An Open-label Multicenter Study on the Efficacy of Continuous Oral Dosing of Vemurafenib on Tumour Response in Previously Treated Patients With Metastatic Melanoma
Brief Title: A Study of Vemurafenib in Previously Treated Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP22657
Record Dates: First submitted 2009-07-28; First posted 2009-07-30 (Estimated); Results first posted 2011-12-22 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Malignant Melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

ARMS (1):
- Single arm (Experimental)
  Interventions: Drug: vemurafenib

INTERVENTIONS:
Drug: vemurafenib — 960 mg b.i.d. continuous oral dosing

SUMMARY:
This open-label single arm study will assess the efficacy, safety and tolerability of Vemurafenib in previously treated patients with metastatic melanoma. Patients will receive oral Vemurafenib [RG7204; PLEXXIKON: PLX4032] at a dose of 960 mg b.i.d. continuously until disease progression or withdrawal from study and will be assessed at regular intervals for tumour response and tolerability. Target sample size is <100 patients.

ELIGIBILITY:
Inclusion Criteria:

* adult patients >/=18 years of age
* histologically confirmed metastatic melanoma (Stage IV, AJCC)
* patients must have completed and failed at least one prior standard of care regimen (e.g. DTIC, temozolomide, etc.)
* BRAF V600E positive mutation (by Roche CoDx BRAF mutation assay)
* measurable disease by RECIST criteria
* negative pregnancy test and, for fertile men and women, effective contraception during treatment and for 6 months after completion

Exclusion Criteria:

* active CNS metastases on CT/MRI within 28 days prior to enrollment
* history of or known carcinomatous meningitis
* previous treatment with BRAF (sorafenib allowed) or MEK inhibitor
* cardiac dysrhythmias >2 NCI CTCAE or treatment with drugs with dysrhythmic potential
* uncontrolled hypertension(>150/100mmHg) despite optimal medical therapy
* infectious disease including HIV, HBV and HCV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2009-09-30 (Actual); Primary Completion 2010-09-27 (Actual); Study Completion 2014-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- United States (12):
  - UCLA - School of Medicine; Division of Hematology/Oncology, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Massachusetts General Hospital;Hematology/ Oncology, Boston, Massachusetts
  - Dana Farber Cancer Inst. ; Dept. of Medical Oncology, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - New York University Medical Center, New York, New York
  - Hospital of the Uni of Pennsylvania; Section of Hematology/Oncology, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt-Ingram Cancer Ctr, Nashville, Tennessee
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Australia (3):
  - Calvary Mater Newcastle; Melanoma Clinic, Newcastle, New South Wales
  - Westmead Hospital; Medical Oncology and Pallative Care, Westmead, New South Wales
  - Peter Maccallum Cancer Institute; Medical Oncology, Melbourne, Victoria

REFERENCES:
- [Derived] Ascierto PA, Ribas A, Larkin J, McArthur GA, Lewis KD, Hauschild A, Flaherty KT, McKenna E, Zhu Q, Mun Y, Dreno B. Impact of initial treatment and prognostic factors on postprogression survival in BRAF-mutated metastatic melanoma treated with dacarbazine or vemurafenib +/- cobimetinib: a pooled analysis of four clinical trials. J Transl Med. 2020 Aug 3;18(1):294. doi: 10.1186/s12967-020-02458-x. PMID 32746839
- [Derived] Frederick DT, Salas Fragomeni RA, Schalck A, Ferreiro-Neira I, Hoff T, Cooper ZA, Haq R, Panka DJ, Kwong LN, Davies MA, Cusack JC, Flaherty KT, Fisher DE, Mier JW, Wargo JA, Sullivan RJ. Clinical profiling of BCL-2 family members in the setting of BRAF inhibition offers a rationale for targeting de novo resistance using BH3 mimetics. PLoS One. 2014 Jul 1;9(7):e101286. doi: 10.1371/journal.pone.0101286. eCollection 2014. PMID 24983357
- [Derived] Lacouture ME, Duvic M, Hauschild A, Prieto VG, Robert C, Schadendorf D, Kim CC, McCormack CJ, Myskowski PL, Spleiss O, Trunzer K, Su F, Nelson B, Nolop KB, Grippo JF, Lee RJ, Klimek MJ, Troy JL, Joe AK. Analysis of dermatologic events in vemurafenib-treated patients with melanoma. Oncologist. 2013;18(3):314-22. doi: 10.1634/theoncologist.2012-0333. Epub 2013 Mar 1. PMID 23457002
- [Derived] Sosman JA, Kim KB, Schuchter L, Gonzalez R, Pavlick AC, Weber JS, McArthur GA, Hutson TE, Moschos SJ, Flaherty KT, Hersey P, Kefford R, Lawrence D, Puzanov I, Lewis KD, Amaravadi RK, Chmielowski B, Lawrence HJ, Shyr Y, Ye F, Li J, Nolop KB, Lee RJ, Joe AK, Ribas A. Survival in BRAF V600-mutant advanced melanoma treated with vemurafenib. N Engl J Med. 2012 Feb 23;366(8):707-14. doi: 10.1056/NEJMoa1112302. PMID 22356324
- [Derived] Su F, Viros A, Milagre C, Trunzer K, Bollag G, Spleiss O, Reis-Filho JS, Kong X, Koya RC, Flaherty KT, Chapman PB, Kim MJ, Hayward R, Martin M, Yang H, Wang Q, Hilton H, Hang JS, Noe J, Lambros M, Geyer F, Dhomen N, Niculescu-Duvaz I, Zambon A, Niculescu-Duvaz D, Preece N, Robert L, Otte NJ, Mok S, Kee D, Ma Y, Zhang C, Habets G, Burton EA, Wong B, Nguyen H, Kockx M, Andries L, Lestini B, Nolop KB, Lee RJ, Joe AK, Troy JL, Gonzalez R, Hutson TE, Puzanov I, Chmielowski B, Springer CJ, McArthur GA, Sosman JA, Lo RS, Ribas A, Marais R. RAS mutations in cutaneous squamous-cell carcinomas in patients treated with BRAF inhibitors. N Engl J Med. 2012 Jan 19;366(3):207-15. doi: 10.1056/NEJMoa1105358. PMID 22256804

RESULTS

PARTICIPANT FLOW:
Groups:
- Vemurafenib 960 mg: Patients received vemurafenib 960 mg (four 240 mg tablets) bid (bis in die, twice daily) orally until disease progression, unacceptable toxicity, withdrawal of consent, or another reason as determined by the investigator.
Period: Overall Study
Arm/Group | Vemurafenib 960 mg
Started | 132
Completed | 84
Not Completed | 48
Not completed — Death | 40
Not completed — Disease progression | 7
Not completed — Withdrawal of consent | 1

BASELINE CHARACTERISTICS:
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.3 (14.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 81

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response (BOR) Assessed by an Independent Review Committee Using Response Evaluation Criteria In Solid Tumors (RECIST 1.1)
Description: BOR was defined as a complete response (CR) or partial response (PR) confirmed per Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. Patients who never received study treatment and treated patients without any post-baseline tumor assessments were considered as non-responders. CR: Disappearance of all target lesions, all non-target lesions, and no new lesion. Any pathological lymph nodes must have had reduction in the short axis to <10 mm. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesion.
Time Frame: From first treatment through September 27, 2010
Population: Intent-to-treat population: All enrolled patients who received at least one, or a partial dose of vemurafenib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 132
Percentage of participants | 52.3 [43.4 to 61.0]

2. Secondary Outcome: Best Overall Response (BOR) Assessed by the Investigator Using Response Evaluation Criteria In Solid Tumors (RECIST 1.1)
Description: as for outcome 1
Time Frame: From first treatment through September 27, 2010
Population: Intent-to-treat population: All enrolled patients who received at least one, or a partial dose of vemurafenib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 132
Percentage of participants | 54.5 [45.7 to 63.2]

3. Secondary Outcome: Duration of Response Assessed by an Independent Review Committee Using Response Evaluation Criteria In Solid Tumors (RECIST 1.1)
Description: Duration of response was defined as the time interval between the date of the earliest qualifying response and the date of disease progression (PD) or death, only for those patients whose best overall response was complete response or partial response. PD: At least 20% increase in the sum of diameters of target lesions compared to Nadir (smallest sum of diameters on-study), unequivocal progression of existing non-target lesions, or presence of new lesion. For patients who were alive without progression, duration of response was censored on the date of the last evaluable tumor assessment.
Time Frame: From first treatment through September 27, 2010
Population: Intent-to-treat population: All enrolled patients who received at least one, or a partial dose of vemurafenib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 69
Months | 6.5 [5.6 to NA] — The upper limit of the confidence interval was not estimable because a large percentage of patients (57%) were progression-free at the data cutoff date and had censored data.

4. Secondary Outcome: Time to Response Assessed by an Independent Review Committee Using Response Evaluation Criteria In Solid Tumors (RECIST 1.1)
Description: Time to response was defined as the interval between the date of the first treatment and the date of the first documentation of confirmed complete response (CR) or partial response (PR), whichever occurred first.
Time Frame: From first treatment through September 27, 2010
Population: Intent-to-treat population: All enrolled patients who received at least one, or a partial dose of vemurafenib.
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 69
Months | 1.38 [1.3 to 1.6]

5. Secondary Outcome: Progression Free Survival (PFS) Assessed by an Independent Review Committee Using Response Evaluation Criteria In Solid Tumors (RECIST 1.1)
Description: PFS was defined the time interval between the date of the first treatment and the date of progression or death from any cause, whichever occurred first. Deaths that occurred in patients without disease progression were considered to be a PFS event on the date of death. Patients who neither progressed nor died were censored on the date of the last evaluable tumor assessment prior to the data cutoff date.
Time Frame: From first treatment through September 27, 2010
Population: Intent-to-treat population: All enrolled patients who received at least one, or a partial dose of vemurafenib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 132
Months | 6.1 [5.5 to 6.9]

6. Secondary Outcome: Overall Survival
Description: Overall survival was defined as the time from the date of the first treatment to the date of death, regardless of the cause of death. For patients who were alive at the time of analysis, overall survival was censored at the last date the patient was known to be alive prior to the data cutoff date.
Time Frame: From first treatment through September 27, 2010
Population: Intent-to-treat population: All enrolled patients who received at least one, or a partial dose of vemurafenib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 132
Months | NA [9.5 to NA] — The median and the upper limit of the confidence interval were not estimable because a large percentage of patients (69%) were alive at the data cutoff date.

7. Secondary Outcome: Improvement in Physical Symptoms (Improvement in Physician's Assessment of Global Performance Status and Oxygen Saturation Requirements, and Decrease in Total Dose and Frequency of Narcotic Pain Analgesics) During Treatment in Comparison to Baseline
Description: Three parameters were measured. (1) Improvement in the Physician's Assessment of Global Performance status on a 7-point scale (1=very much better to 7=very much worse). (2) Improvement in oxygen saturation requirements, defined as a clinically meaningful increase in oxygen saturation requirement (from a baseline value < 95% to ≥ 95% saturation using a pulse oximeter). (3) A decrease in total dose and frequency of narcotic pain analgesics. The percentage of patients showing improvement (1 and 2) or a decrease (3) are reported.
Time Frame: From first treatment through September 27, 2010
Population: Intent-to-treat population: All enrolled patients who received at least one, or a partial dose of vemurafenib.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 132
Percentage of participants
  Improvement in performance status | 83.3 [80.0 to 90.0]
  Improvement in oxygen saturation requirement | 4.5 [0.0 to 10.0]
  Decrease in use of narcotic pain analgesics | 3.0 [0.0 to 10.0]

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Vemurafenib on Day 15 of Cycle 1
Description: Blood samples for assessing the concentration of vemurafenib in plasma were drawn before the morning dose and at 2, 4, 6, and 8 hours post-dose on Day 15 of Cycle 1. Pharmacokinetic parameters were estimated by non-compartmental analysis (Win Non-Lin).
Time Frame: Pre-dose to 8 hours post-dose on Day 15 of Cycle 1
Population: Pharmacokinetic population: All patients who received all doses of vemurafenib without dose reduction up to and including Day 15 and who provided at least one of the pharmacokinetic assessments up to and including 8 hours after the first daily dose on Day 15.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 87
μg/mL | 56.73 (21.76)

9. Secondary Outcome: Vemurafenib Plasma Level Area Under the Curve From 0 to 8 Hours (AUC0-8h) on Day 15 of Cycle 1
Description: Blood samples for assessing the concentration of vemurafenib in plasma were drawn before the morning dose and at 2, 4, 6, and 8 hours post-dose on Day 15 of Cycle 1. Pharmacokinetic parameters were estimated by non-compartmental analysis (Win Non-Lin). AUC0-8h was calculated using the linear trapezoidal rule.
Time Frame: Pre-dose to 8 hours post-dose on Day 15 of Cycle 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg⋅h/mL
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 87
μg⋅h/mL | 380.16 (143.56)

10. Secondary Outcome: Vemurafenib Plasma Levels at Various Treatment Cycles
Description: Blood samples for assessing the concentration of vemurafenib in plasma were drawn before the morning dose and 4 hours post-dose at Day 1 of Cycles 1, 2, 3, 4, 6, 8, and 10. Each Cycle was 3 weeks in duration.
Time Frame: Pre-dose Cycle 1 Day 1 to 4 hours post-dose Cycle 10 Day 1
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 122
μg/mL
  Pre-dose Cycle 1 Day 15, n=108 | 47.55 (23.14)
  Pre-dose Cycle 2 Day 1, n=122 | 41.12 (23.39)
  Pre-dose Cycle 3 Day 1, n=109 | 45.20 (21.33)
  Pre-dose Cycle 4 Day 1, n=109 | 50.31 (19.52)
  Pre-dose Cycle 6 Day 1, n=96 | 50.38 (19.54)
  Pre-dose Cycle 8 Day 1, n=71 | 50.42 (22.06)
  Pre-dose Cycle 10 Day 1, n=50 | 50.78 (20.19)
  4 hours post-dose Cycle 2 Day 22, n=93 | 48.38 (20.00)
  4 hours post-dose Cycle 3 Day 43, n=78 | 50.79 (19.20)
  4 hours post-dose Cycle 4 Day 1, n=75 | 55.76 (20.57)
  4 hours post-dose Cycle 6 Day 1, n=58 | 58.92 (20.12)
  4 hours post-dose Cycle 8 Day 1, n=43 | 58.95 (20.98)
  4 hours post-dose Cycle 10 Day 1, n=27 | 63.27 (21.52)

11. Secondary Outcome: Time-matched Change From Baseline in the Study Specific Corrected QT Interval (QTcP)
Description: Three electrocardiograms (ECG) were obtained pre-dose and 2, 4, 6, and 8 hours post-dose at Days 1 and 15 of Cycle 1 and again pre-dose and 4 hours post-dose at various Cycles throughout treatment. Five baseline triplicate ECGs were obtained before the start of treatment at the same time points used during treatment. Reported is the largest mean time-matched QTcP change from baseline. QTcP=QT/(60/heart rate)^β (β=mean [calculated separately for males and females] log-transformed QT versus log-transformed RR regression slopes using all available pre-treatment (baseline) ECG values.
Time Frame: Pre-dose Cycle 1 Day 1 to pre-dose Cycle 6 Day 1
Population: Electrocardiogram (ECG) evaluable population: All treated patients who had a baseline ECG and at least one ECG during treatment.
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 128
ms
  Cycle 1 Day 15 at 2 hours post-dose, n=109 | 12.8 [NA to 14.9] — This is a one-sided confidence interval.
  Cycle 6 Day 1 at pre-dose, n=85 | 15.1 [NA to 17.7] — This is a one-sided confidence interval.

12. Secondary Outcome: Percentage of Patients With Adverse Event
Description: The intensity of adverse events was graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events v 4.0 (CTCAE) on a 5-point scale (Grade 1 to 5: Mild, Moderate, Severe, Life-threatening, and Death).
Time Frame: From first treatment through September 27, 2010
Population: Intent-to-treat population: All enrolled patients who received at least one, or a partial dose of vemurafenib.
Measure: Number; unit: Percentage of participants
Arm/Group | Vemurafenib 960 mg
Number analyzed (Participants) | 132
Percentage of participants | 100.0

ADVERSE EVENTS:
Time Frame: Screening through 6 months after the last patient enrolled
Arm/Group | Vemurafenib 960 mg
Serious Adverse Events (participants affected / at risk) | 67/132
Other Adverse Events (participants affected / at risk) | 131/132
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib 960 mg (N=132)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 28
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
DYSPHAGIA (Gastrointestinal disorders) | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 2
NAUSEA (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
DIARRHOEA (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
OESOPHAGITIS (Gastrointestinal disorders) | 1
PANCREATITIS (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
PNEUMONIA (Infections and infestations) | 3
CELLULITIS (Infections and infestations) | 2
BREAST CELLULITIS (Infections and infestations) | 1
PSEUDOMONAS INFECTION (Infections and infestations) | 1
SALMONELLOSIS (Infections and infestations) | 1
SKIN INFECTION (Infections and infestations) | 1
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 1
WOUND INFECTION (Infections and infestations) | 1
CONVULSION (Nervous system disorders) | 3
FACIAL PALSY (Nervous system disorders) | 3
PYREXIA (General disorders) | 3
MULTI-ORGAN FAILURE (General disorders) | 1
PAIN (General disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 3
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 2
BLOOD BILIRUBIN INCREASED (Investigations) | 2
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1
BILIRUBIN CONJUGATED INCREASED (Investigations) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 2
ANGINA PECTORIS (Cardiac disorders) | 1
PERICARDITIS (Cardiac disorders) | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1
HEPATIC CYST (Hepatobiliary disorders) | 1
JAUNDICE (Hepatobiliary disorders) | 1
DEHYDRATION (Metabolism and nutrition disorders) | 2
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 1
EXFOLIATIVE RASH (Skin and subcutaneous tissue disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 1
RASH VESICULAR (Skin and subcutaneous tissue disorders) | 1
DELIRIUM (Psychiatric disorders) | 1
PSYCHOTIC DISORDER (Psychiatric disorders) | 1
RENAL FAILURE (Renal and urinary disorders) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
ANAEMIA (Blood and lymphatic system disorders) | 1
RETINAL VEIN OCCLUSION (Eye disorders) | 1
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
DEEP VEIN THROMBOSIS (Vascular disorders) | 1
ATRIAL FLUTTER (Cardiac disorders) | 1
LEFT LUNG GROUND GLASS OPACITIES-PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vemurafenib 960 mg (N=132)
RASH (Skin and subcutaneous tissue disorders) | 68
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 65
ALOPECIA (Skin and subcutaneous tissue disorders) | 47
PRURITUS (Skin and subcutaneous tissue disorders) | 40
SKIN PAPILLOMA (Skin and subcutaneous tissue disorders) | 39
HYPERKERATOSIS (Skin and subcutaneous tissue disorders) | 37
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 27
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 22
DRY SKIN (Skin and subcutaneous tissue disorders) | 21
RASH PAPULAR (Skin and subcutaneous tissue disorders) | 17
KERATOSIS PILARIS (Skin and subcutaneous tissue disorders) | 12
ERYTHEMA (Skin and subcutaneous tissue disorders) | 11
PALMAR-PLANTAR (Skin and subcutaneous tissue disorders) | 11
ERYTHRODYSAESTHESIA SYNDROME ACNE (Skin and subcutaneous tissue disorders) | 10
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 9
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 8
SKIN LESION (Skin and subcutaneous tissue disorders) | 8
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 86
MYALGIA (Musculoskeletal and connective tissue disorders) | 31
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 15
BACK PAIN (Musculoskeletal and connective tissue disorders) | 14
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 12
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 12
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 7
FATIGUE (General disorders) | 71
OEDEMA PERIPHERAL (General disorders) | 30
PYREXIA (General disorders) | 20
CHILLS (General disorders) | 9
PAIN (General disorders) | 7
VISION BLURRED (Eye disorders) | 7
NAUSEA (Gastrointestinal disorders) | 47
DIARRHOEA (Gastrointestinal disorders) | 37
VOMITING (Gastrointestinal disorders) | 33
CONSTIPATION (Gastrointestinal disorders) | 21
ABDOMINAL PAIN (Gastrointestinal disorders) | 12
DYSPEPSIA (Gastrointestinal disorders) | 11
DECREASED APPETITE (Metabolism and nutrition disorders) | 28
HEADACHE (Nervous system disorders) | 36
DYSGEUSIA (Nervous system disorders) | 14
NEUROPATHY PERIPHERAL (Nervous system disorders) | 13
DIZZINESS (Nervous system disorders) | 8
HYPOKALAEMIA (Metabolism and nutrition disorders) | 10
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 7
SUNBURN (Injury, poisoning and procedural complications) | 19
COUGH (Respiratory, thoracic and mediastinal disorders) | 16
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 13
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 10
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 17
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 10
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 8
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 7
BLOOD CREATININE INCREASED (Investigations) | 12
LYMPHOCYTE COUNT DECREASED (Investigations) | 7
SEBORRHOEIC KERATOSIS (Skin and subcutaneous tissue disorders) | 19
FOLLICULITIS (Infections and infestations) | 12
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 8
NASOPHARYNGITIS (Infections and infestations) | 7
BLOOD BILIRUBIN INCREASED (Investigations) | 7
WEIGHT DECREASED (Investigations) | 12
ANAEMIA (Blood and lymphatic system disorders) | 11
DEPRESSION (Psychiatric disorders) | 11
INSOMNIA (Psychiatric disorders) | 9
ANXIETY (Psychiatric disorders) | 7
ACNE (Skin and subcutaneous tissue disorders) | 10
MELANOCYTIC NAEVUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.